CLINICAL TRIAL: NCT06091631
Title: Effect of Magnesium Sulfate Nebulization on Postoperative Sore Throat and Stress Response Induced Tracheal Intubation
Brief Title: Magnesium Sulfate in Surgical Stress Attenuation Postoperative Sore Throat and Stress Response Induced Tracheal Intubation
Acronym: Magnesium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayman Abd El-Khalek Mohammed Glala, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Attenuation of surgical stress
Record Dates: First submitted 2023-10-02; First posted 2023-10-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Anesthesia Complication; Anesthesia Intubation Complication
Keywords: Magnesium sulfate; anesthesia stress response for intubation

STUDY DESIGN:
Intervention Model Description: 2 groups are investigated. Each group consists of 50 patients. First group will receive magnesium sulfate inhalation . The other group will receive distilled water inhation
Who Masked: Participant
Masking Description: the participant will not know whither a magnesium sulfate inhalation or distilled water in the vaporizer
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium sulfate (Experimental): will receive magnesium sulfate inhation
  Interventions: Procedure: Magnesium sulfate vaporization
- Control (No Intervention): Will receive distilled water vaporization

INTERVENTIONS:
Procedure: Magnesium sulfate vaporization — pre-opeative magnesium sulfate vaporization
  Arms: Magnesium sulfate

SUMMARY:
Magnesium sulfate has many mechanisms of action for attenuating the stress response as inhibition of catecholamine releasing from the adrenal medulla, keeping the plasma concentration of epinephrine at a fixed level, decreasing the circulating norepinephrine level when compared to that of a control group[ and also has a vasodilation effect on systemic and coronary blood vessels by blocking calcium ion in vascular smooth muscle.-Methyl- D-Aspartate (NMDA) antagonism is an amazing recent discovery for magnesium sulphate to play an important role in stress response.

In this study, we will study the effects of nebulized magnesium sulfate on hemodynamics during intubation.

DETAILED DESCRIPTION:
Inclusion criteria

* 20-50 years old
* ASA: 1, 2
* Elective fit laparoscopic cholecystectomy Exclusion criteria
* Patient refusal
* patients with history of hypersensitivity to magnesium sulphate
* patients with coronary ischemic disease, atrioventricular block of any degree, known cardiac arrhythmias, heart failure
* on beta blockers or calcium channel blockers
* expected difficult intubation (Mallampati 4)
* Body mass index > 40

Study tools:

Following institutional ethical committee approval and written informed consent,a prospective randomized double-blinded study. After written informed consent wil be given, 100 patients, ASA 1 or 2, aged between 20 - 50 years, scheduled for elective surgery with Orotracheal Intubation (OTI) will be assessed for eligibility. Patients will be recruited in the study divided into two equal groups; Patients in Group A: will receive nebulized magnesium sulfate in 3 ml (240 mg) over 15 min, While group B: will receive nebulized normal saline in 3 ml over 15 min, ending 5 min before the induction of anesthesia. SBP, DBP, HR, and blood glucose level will be measured at the following intervals; Baseline (before induction), after premedication (sedation), after induction, after ETT intubation, 3 min later, 6 min later.

Full monitoring data (Blood pressure every 3 minutes, ECG, Nanogram, and pulse oximeter) wil be collected till 6 minutes then every 5 minutes. Random blood sugar will be tested 5 minutes pre-intubation, 3minutes and 5 minutes after intubation.

After end of nebulization, sedation with 2 mg midazolam and IV fluids (10 ml/kg) will be infused to avoid tachycardia of dehydration and fear of surgery. Then, we proceed on general anesthesia through propool titration + fentanyl 100 mcg + Cisatracurium 0.15 mg/kg. Endotracheal intubation with cuffed tube and mechanical ventilation with mild increase in respiratory rate 14-16/min to overcome CO2 peritoneal insufflation. All patients will receive intraoperatively, nalbuphine 0.1 mg/kg + ketorolac 60 mg + paracetamol IV 1 g. Dexamethasone 4mg + Ondansetron 4mg will be received to all patients for prophylaxis against postoperative nausea and vomiting. After end of surgery, cessation of inhalational anesthesia and reversal of muscle relaxation with neostigmine 2.5 mg+ Atropine 1mg will be done.

Consumption of isoflurane intraoperatively will be recorded. Post operative assessment for pain using VAS score will be assessed 2 hours after recovery.

Time for recovery after stop of isoflurane will be estimated.

ELIGIBILITY:
Inclusion Criteria:

* 20-50 years old
* ASA: 1, 2
* Elective fit laparoscopic cholecystectomy

Exclusion Criteria:

* -Patient refusal
* patients with history of hypersensitivity to magnesium sulphate
* patients with coronary ischemic disease, atrioventricular block of any degree, known cardiac arrhythmias, heart failure
* on beta blockers or calcium channel blockers
* expected difficult intubation (Mallampati 4)
* Body mass index > 40

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of post-operative sore throat at 0 hours in both groups | at 0 hours in both groups
  Incidence of post-operative sore throat 0 h
Incidence of post-operative sore throat at 2 hours in both groups | at 2 hours in both groups
  Incidence of post-operative sore throat 2 h
Incidence of post-operative sore throat at 4 hours in both groups | at 4 hours in both groups
  Incidence of post-operative sore throat 4 h
Incidence of post-operative sore throat at 24 hours in both groups | at 24 hours in both groups
  Incidence of post-operative sore throat 24 h

SECONDARY OUTCOMES:
Improvement in postoperative stress response after (3, 6) minutes including: • Heart rate > 20% baseline • Systolic and mean BP >25% baseline • Random blood sugar increase > 50 mg/dl from baseline | (3, 6) minutes
  Improvement in postoperative stress response after (3, 6) minutes including:
  * Heart rate > 20% baseline
  * Systolic and mean BP >25% baseline
  * Random blood sugar increase > 50 mg/dl from baseline
Effect on Pain score VAS 2hours after recovery | 2hours after recovery
  Effect on Pain score VAS visual analogue scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, faculty of medicine, anesthesia and ICU and pain management department, Asyut, Asyut Governorate, Egypt